CLINICAL TRIAL: NCT02055989
Title: A Phase I/II Study of the Use of Intensity Modulated Radiotherapy (IMRT) in Cancer of the Thyroid, Larynx and Hypopharynx
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 1978
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Locally Advanced Larynx, Hypopharyngeal Squamous Cell Cancers; Locally Advanced Thyroid Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-escalated radiotherapy level 1 (Experimental)
  Interventions: Radiation: Dose-escalated radiotherapy level 1
- Sequential dose-escalated radiotherapy level 2 (Experimental)
  Interventions: Radiation: Sequential dose-escalated radiotherapy level 2

INTERVENTIONS:
Radiation: Dose-escalated radiotherapy level 1
  Arms: Dose-escalated radiotherapy level 1
Radiation: Sequential dose-escalated radiotherapy level 2
  Arms: Sequential dose-escalated radiotherapy level 2

SUMMARY:
This study is a phase I/II dose escalation trial designed to test the feasibility of delivering IMRT to thyroid, larynx and hypopharynx cancer patients, and to assess the safety and possible improvement in outcome when the dose is increased.

This protocol is in fact two studies running in parallel: thyroid cancer patients and larynx/ hypopharynx cancer patients. These two groups of patients are being treated differently and will be analysed separately.

The primary objective of this Phase I sequential cohort study was to determine the feasibility of delivering modest acceleration and dose-escalated IMRT in locally advanced high-risk thyroid cancers. We report the incidence and prevalence of acute toxicities of 2 dose fractionation regimens.

DL1: primary site 58.8 Gy in 28 daily fractions and nodal levels 50 Gy in 28 daily fractions

DL2: primary 66.6 Gy in 30 daily fractions and post operative nodal levels 60 Gy in 30 daily fractions and elective nodal levels 54 Gy in 30 daily fractions

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically confirmed squamous cell or undifferentiated carcinoma of the head and neck.
2. Newly diagnosed histologically confirmed papillary,follicular, undifferentiated or medullary carcinoma of the thyroid.
3. Tumours arising from the oral larynx or hypopharynx requiring radical radiation of the primary tumour by parallel opposed lateral fields, and bilateral cervical lymph node irradiation.
4. High risk of radiation induced xerostomia with conventional radiotherapy due to the irradiation of the majority of both parotid glands (defined as estimated mean dose to both parotid glands greater than 26 Gy using conventional radiotherapy technique).
5. Radiotherapy either as primary therapy or post-operative (only for thyroid carcinoma). Techniques to be detailed by each centre. Neo-adjuvant and concomitant chemotherapy are permitted.
6. Stage T1-4, N1-3, M0 disease
7. Zubrod Performance Status 0-2

Exclusion Criteria:

1. Previous radiotherapy to the head and neck region
2. Previous malignancy except non-melanoma skin cancer
3. Previous or concurrent illness which in the investigators opinion would interfere with either completion of therapy or follow-up
4. Prophylactic use of amifostine or pilocarpine is not allowed
5. Brachytherapy is not allowed as part of the treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2002-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of patients with grade 3 or 4 complication at 12 months after treatment. | 12 months after radiotherapy

SECONDARY OUTCOMES:
Acute toxicity | Up to 3 months after radiotheapy
Late toxicity | Up to 60 months after radiotherapy
Local control | Up to 60 months after radiotherapy
Loco-regional control | Up to 60 months after radiotherapy
Loco-regional disease free survival (disease free thyroid bed, neck and superior mediastinum) | Up to 60 months after radiotherapy
Disease free survival | Up to 60 months after radiotherapy
Overall Survival | Up to 60 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Chris M Nutting, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, London, United Kingdom